CLINICAL TRIAL: NCT03126760
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Parallel Group, Pilot Study to Assess the Efficacy and Safety of Acthar® in Subjects With Relapsing-remitting Multiple Sclerosis
Brief Title: Acthar Gel for Multiple Sclerosis That Keeps Getting Better and Worse (RRMS)
Acronym: OPTIONS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment difficulties and COVID-19 logistical challenges; no safety concerns
Sponsor: Mallinckrodt ARD LLC (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MNK14274069
Record Dates: First submitted 2017-04-04; First posted 2017-04-24 (Actual); Results first posted 2021-06-03 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Relapsing, Remitting Multiple Sclerosis; RRMS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: While Care Provider and Outcomes Assessor were also blinded, it was considered a double-blind study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acthar Gel (Experimental): Participants receive Acthar Gel under the skin once a day for 14 consecutive days
  Interventions: Drug: Acthar Gel
- Placebo (Placebo Comparator): Participants receive Placebo under the skin once a day for 14 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acthar Gel — Acthar Gel 1 mL (80U) for subcutaneous injection
  Other Names: Repository Corticotropin Injection
  Arms: Acthar Gel
Drug: Placebo — Placebo for subcutaneous injection
  Other Names: Matching Placebo
  Arms: Placebo

SUMMARY:
This study will enroll about 66 participants who experienced a relapse of RRMS that steroids did not help. The doctor will put participants into a treatment group. Each person has an equal chance of being in either one of two groups (like flipping a coin). One group will receive a shot of study medicine (called Acthar Gel) under their skin every day for 14 days. The other group will receive a shot every day for 14 days, too, but there is no medicine in it (called placebo).

ELIGIBILITY:
Key Inclusion Criteria:

* Had a clinical diagnosis of relapsing-remitting multiple sclerosis (RRMS)
* Had a relapse with onset ≤42 days prior to the Baseline Visit
* Had started treatment with 3 to 5 days (inclusive, over a period of up to 7 days) of specific high dose corticosteroids within 28 days of the onset of the first relapse symptom
* Had failed to obtain improvement of at least 1 point in one or more functions on the Function Systems Score (FSS) 14 days following their first dose of high dose corticosteroids
* Has an Expanded Disability Index Scale (EDSS) score of 2.0 to 6.5 (inclusive) at the Baseline Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (22):
- United States (22):
  - Stanford University Medical Center, Palo Alto, California
  - Advanced Neurosciences Research LLC, Fort Collins, Colorado
  - University of South Florida, Bradenton, Florida
  - Neurology Associates, P. A., Maitland, Florida
  - University of Miami - Miller School of Medicine, Miami, Florida
  - Tallahassee Neurological Clinic, PA, Tallahassee, Florida
  - Multiple Sclerosis Center of Atlanta, Atlanta, Georgia
  - Meridian Clinical Research LLC, Savannah, Georgia
  - Consultants in Neurology LTD, Northbrook, Illinois
  - OSF Healthcare System Saint Francis Medical Center, Peoria, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Wayne State University (WSU) - Multiple Sclerosis Treatment and Clinical Research Center (MS Center), Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - University of Buffalo, Buffalo, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Cincinnati Physicians Company, LLC, Dayton, Ohio
  - Northern Ohio Neuroscience, LLC, Sandusky, Ohio
  - Texas Neurology, PA, Dallas, Texas
  - Neurology Center of San Antonio, San Antonio, Texas
  - MultiCare Neuroscience Center of WA, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No
Discussion of statistical endpoints and analysis are included in manuscripts. Summary aggregate (basic) results (including adverse events information) and the study protocol are made available on clinicaltrials.gov (NCT03126760) when required by regulation. Individual de-identified patient data will not be disclosed. Requests for additional information should be directed to the company at medinfo@mnk.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated early by sponsor decision because of recruitment difficulties and the impact of the COVID-19 pandemic.
Pre-assignment Details: Approximately 66 participants were planned at 25 sites; while only 35 were randomized using 31 sites, because of recruitment difficulties and the impact of the COVID-19 pandemic.
Period: Overall Study
Arm/Group | Acthar Gel | Placebo
Started | 18 | 17
Modified Intent to Treat (mITT) (All participants who received study treatment) | 18 | 17
Completed Treatment | 17 (One participant halted treatment for adverse event, but completed the study) | 17
Completed | 18 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Acthar Gel | Placebo | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Median (Full Range); unit: years] | 40 [21 to 62] | 43 [26 to 64] | 40 [21 to 64]
Age, Customized [Count of Participants; unit: Participants]
  Adults 21-64: ≤35 | 4 | 6 | 10
  Adults 21-64: 36-45 | 10 | 6 | 16
  Adults 21-64: 46-55 | 2 | 2 | 4
  Adults 21-64: 56-64 | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 17 | 16 | 33
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Score on the Expanded Disability Status Scale (EDSS) at Baseline and Day 42
Description: The EDSS is a 10-point assessment of neurological impairment/disability in multiple sclerosis (MS) patients, ranging from 0 (normal neurological examination) to 10 (death due to MS). EDSS is rated by a person who only collects outcome measures, and has no knowledge of the treatment received.
Time Frame: Baseline, Day 42
Population: modified Intent to Treat (mITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acthar Gel | Placebo
Number analyzed (Participants) | 18 | 17
score on a scale
  Baseline | 3.86 (1.122) | 3.85 (1.169)
  Day 42 | 2.92 (0.974) | 3.62 (1.485)

ADVERSE EVENTS:
Time Frame: 42 days
Description: Treatment emergent serious and non-serious adverse events are recorded. Treatment emergent is defined as adverse events that started or worsened in severity on or after the first dose of study drug. Clinically significant change in vital signs, laboratory values and/or physical examinations are recorded as adverse events.
Arm/Group | Acthar Gel | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 14/18 | 12/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acthar Gel (N=18) | Placebo (N=17)
Goitre (Endocrine disorders) | 0 | 1
Corneal degeneration (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Feeling jittery (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Injection site bruising (General disorders) | 3 | 4
Injection site discomfort (General disorders) | 0 | 1
Injection site erythema (General disorders) | 1 | 2
Injection site haemorrhage (General disorders) | 1 | 0
Injection site inflammation (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Injection site reaction (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Heart rate increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Protein total decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Plica syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early by sponsor decision because of recruitment difficulties and the impact of the COVID-19 pandemic. The planned analyses did not change except that the total sample size was reduced. Inferential statistics were not performed. Results are nominal because the sample size did not reach that specified in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT03126760/Prot_SAP_001.pdf